CLINICAL TRIAL: NCT05646160
Title: Effects of Myofascial Trigger Points Therapy in Migraine.
Brief Title: Effects of MTRPs Therapy in Migraine.
Acronym: MTRPs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Józef Piłsudski University of Physical Education (Other)
Collaborators: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Maciej Olesiejuk, Principal Investigator, PhD, Józef Piłsudski University of Physical Education
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKE 01-52 / 2017; 14/21//10/11/2017 (Registry Identifier: Regional Research and Development Center in Biała Podlaska)
Record Dates: First submitted 2022-11-23; First posted 2022-12-12 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Migraine; Pain, Shoulder; Trapezius Muscle Strain Left; Trapezius Muscle Strain Right; Muscle Pain; Trigger Point Pain, Myofascial; Cervical Pain
Keywords: myometrics; range of motion; migraine; blood tests; muscle pain; ischemic compression Myofascial Trigger Points (IC-MTRPs); muscle mechanical properties
MeSH Terms: conditions — Migraine Disorders; Shoulder Pain; Myalgia; Myofascial Pain Syndromes; Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- chronic migraine (CM) (Experimental): CM is diagnosed after a patient has experienced a tension or migraine headache for at least 15 days in a month for at least 3 months, when not less than 8 days is characterized by the symptoms typical of migraine diagnosis.
  Interventions: Other: Ischemic Compression of Myofascial Trigger Points (IC-MTRPs)
- episodic migraine with aura (EMa) (Experimental): EMa, known as classical migraine, is characterized by an attack of pain lasting several or tens of minutes, during which the appearance of unilateral visual and sensory symptoms from the central nervous system, usually associated with pain and migraine symptoms.
  Interventions: Other: Ischemic Compression of Myofascial Trigger Points (IC-MTRPs)
- episodic migraine without aura (EMb) (Experimental): EMb is diagnosed after at least 5 attacks per month, characterized by a one-sided, pulsating headache of moderate or severe intensity, which increases with physical activity, sometimes with vomiting, and sensitivity to light and sound. This episode of migraine must last from 4 to 72 hours.
  Interventions: Other: Ischemic Compression of Myofascial Trigger Points (IC-MTRPs)

INTERVENTIONS:
Other: Ischemic Compression of Myofascial Trigger Points (IC-MTRPs) — IC-MTrPs intervention was made first on the right side and then on the left side and this order was the same in each patient. Before starting the therapeutic procedure, the MTrPs localizations were identified by palpation and pinch pressure in patients lying back on the couch. During the procedure, a qualified physiotherapist sat behind the subject's head. The pressure was sustained for about 5 seconds with a 2-3 seconds pause. In each subject, the intervention lasted 15 minutes on the same measurement day in the morning. The subjects underwent cycle of seven IC-MTrPs therapeutic sessions, with 3 days brakes between each session, that lasted in total about a 3-weeks (25 days).
  Other Names: MTRPs therapy; trigger points therapy/compression

SUMMARY:
Case series, repeated-measures design, pilot study.

Adult, female, migraine patients underwent seven Ischemic Compression Myofascial Trigger Points (IC-MTrPs) therapy sessions.

The aim of the study is to investigate whether therapy of the shoulder girdle and neck muscles by deactivating MTrPs causes modification of biomechanical and biochemical variables in the blood and reduces headache in people with migraine, improving their quality of life by improving their health.

People qualified for the study were divided into 3 groups according to the type of migraine:

1. CM group - patients with chronic migraine
2. EMa group - patients with paroxysmal migraine with aura
3. EMb group - patients with paroxysmal migraine without an aura.

All patients underwent 7 interventions in the area of the muscles of the shoulder girdle and neck (by deactivating trigger points) performed every 2 or 3 days. They did not take any headache medications during the treatment period. However, during a migraine attack, they could undergo treatments and research measurements. Biomechanical measurements of the cervical spine, shoulder girdle muscles and blood chemistry were performed before, during and after the patients' therapy.

All treatments were performed on the following muscles:

* m. trapesius pars descendent (trapezius upper),
* m. sternocleidomastoideus (sternocleidomastoid),
* m. temporalis (temporal),
* m. legator scapulae (levator scapula),
* m. supraspinatus (supraspinatus),
* m. suboccipitales (suboccipital).

DETAILED DESCRIPTION:
Detailed Description:

I. The specific objectives were to investigate whether the therapy of the shoulder girdle and neck had an effect on:

1. the range of mobility of the cervical spine
2. myometric variables (stiffness, flexibility and tension) of the muscle (trapezius upper part)
3. concentration of selected biochemical factors (S100 beta protein, substance P (SP), calcitonin gene-related peptide (CGRP), brain-derived neurotrophic factor (BDNF) in patients with migraine
4. feel headache
5. feel pain in the muscles of the shoulder girdle
6. feel the quality of life related to health.

II. Hypotheses

1. Inactivation of MTrPs by IC-MTRPs therapy improves biomechanical properties of the cervical spine (increases the range of mobility of the cervical spine - lateral inclination, rotation and forward inclination) in people with migraine.
2. Inactivation of MTrPs by IC-MTRPs therapy improves the resting biomechanical properties (reduction of tension, stiffness and increased flexibility) of the muscles of the shoulder girdle.
3. Inactivation of MTrPs by IC-MTRPs therapy reduces the concentration of biochemicals in the blood responsible for the aggravation of migraine pain.
4. TOBS therapy through IC-MTrPs therapy improves biomechanical and biochemical variables, reducing the sensations of headache and muscle pain, improving health-related quality of life in people with migraine.

III. The course of research. Before and during the intervention cycle, migraine patients were subjected to biomechanical and biochemical tests. In the morning, fasting blood was drawn on the first and last day of therapy, before and after the intervention, in order to determine the biochemical parameters. Before the start of therapy and one month after the last intervention, the patients completed the WHOQoL-BREF (WHO Quality of Life BREEF) and the VAS (visual analogue scale) for headache and muscle pain during therapy. Before and after the first, fourth and seventh interventions, and one month after the last treatment, myometric measurements of muscle tension, stiffness and flexibility were performed using the Myoton Pro 3 apparatus (Tallinn, Estonia), and biomechanical measurements of cervical spine mobility using the Myo Motion apparatus (Noraxon, Scottsdale, USA). Muscle pain and headache during the procedure were also assessed using the VAS scale.

The research was carried out during eight research sessions in the morning, which were carried out according to a strictly defined scheme (for all subjects in the same order and location)

IV. Research methods. IV (I) Anthropometric measurements. The subjects' height, weight and body composition were measured using the Tanita BC 418 ma electronic system (Tanita Corporation, Tokyo, Japan T174). Measurement of body mass composition was determined by the electrical bioimpedance (BIA) method. The obtained data were necessary to carry out myometric and accelerometric measurements (mobility of the cervical spine), where it was required to provide the current weight and height of the examined person.

IV (II) Biochemical determinations. Blood collection and serum collection. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am before and after the treatment on the first day and 24 hours after the sixth treatment, into test tubes without serum anticoagulants. The sterile blood (8 ml) was left for 30 min at room temperature, then the blood was centrifuged at 1500 rpm / min x g for 10 min. Serum was transferred to new 300 µl tubes and stored at -70 ° C until biochemical determinations were made.

Determination of the concentration of SP and S100B, CGRP, BNDF with the immunochemical method of ELISA The concentration of substance P, protein S100beta, calcitonin gene-related peptide (CGRP), BNDF (brain-derived neurotrophic factor) was determined using the immunochemical ELISA method in accordance with the instructions of the kit manufacturers (R&D systems, Londyn UK).

IV (III) Biomechanical measurements of the cervical spine Determination of biomechanical parameters of the cervical spine. For mobility measurements, a set for recording and analyzing human movement in 3D with the use of Noraxon Myo Motion accelerometric sensors (Noraxon, Scottsdale, USA) was used. The measuring device allowed to assess the range of movement of the cervical spine with the motor control of the patient in the movement of the lateral to the right bend and left side, right and left rotations and forward bends. Automatic recording of motion parameters completely eliminated errors related to the subjective assessment of a diagnostician with the use of manual measuring tools. The ROM values will be expressed in degrees [°].

Sensors (sensor 1 was mounted at the height of the first spinous process of the thoracic spine (Th1), sensor 2 was mounted on the occiput (Co)) mounted on the patient's head, on an elastic band, have the function of automatic, wireless calibration, thanks to which the above-described data was collected before and after day 1, 4 and 7 of therapy for the muscles of the shoulder girdle and neck and for 1 month after the last intervention. Each of the examined women sat on a stiff armchair, fastened with belts preventing the movement of the torso in order to eliminate measurement errors resulting from the human factor. The examined person made a given neck movement at the clear command of the researcher. First left side bend, then right side bend, then left head rotation, then right side bend, last head tilt forward. The range of motion measured in the research was expressed in degrees. The examiner carried out the measurements without knowing about the study group (blinding) and did not participate in the analysis of the obtained data.

IV (IV) Myometric measurements of the muscle properties of the shoulder girdle (tension, stiffness and flexibility) of the muscles.

The muscle properties were tested using a Myoton Pro 3 miometer (Myoton, Tallinn, Estonia). The measurement is non-invasive and fast, it takes from 3 to 30 seconds depending on the selected option. In the presented work, the 10 measurement repetition mode was selected, from which the device software calculated the average for each of the three parameters (tension, stiffness and elasticity) and saved it in the device memory. The measurement consisted in placing the measuring tip of the myometer always perpendicular to the skin surface at a strictly defined point before and after the therapy. The researcher moved the device towards the examined tissue until the green light on the body of the device turned on. Such an operation activates the electromagnetic mechanism, which generated mechanical impulses with a constant force deforming the muscle at the measuring point through the moved measuring tip. The meter automatically performed a series of pulses (10), and the researcher held the device steadily in the selected position. The pressure of the tip (punch) is short (10 ms) and of low force (0.40 N), which does not cause a neurological reflex muscle contraction response. The impulse caused mechanical vibrations of the examined muscle, according to which the following parameters were calculated after automatic processing by the accelerometric recording processor:

* F (frequency) - it determines the muscle tension and is calculated as the maximum frequency from the power of the accelerometric signal spectrum and is expressed as in hertz [Hz].
* S (stiffness) - is calculated from the formula S-MYO = amax. mprobe / ^ l, where amax is the maximum acceleration of the striking measuring tip [kg], a ^ l is the maximum distance the stylus has moved [m]. This parameter is expressed in [N / m] and determines the force generated by the measuring tip of the myometer needed to deform the tested tissue to a specific depth.
* D (decrement) - free decrease of vibration calculated from the logarithm:

Patient seated steadily and relaxed in a chair with full body support, hands in lap, looking straight ahead. For all patients, six measurement points were carefully indicated on both sides of upper trapezius muscle, i.e. three points on the left upper trapezius (P1, P2, P3) and three on the right upper trapezius (P4, P5, P6). The three testing points were located on an horizontal line between the cervico-thoracic junction of the spine (C7 / Th1) and the shoulder process of scapula in a distance between these points similar for each patient. Going from medial to lateral side the testing points were as follows: (i) the most medial point as P1 on the left and P4 on the right trapezius, which was distant 3 cm laterally from the cervico-thoracic junction of the spine (C7 / Th1); (ii) the next P2 or P5 point (intermediate one) was distant 2 cm laterally from the P1 or P4; (iii) and the most laterally located the P3 or P6 point was distant 2 cm from the P2 or P5 (on the left or right trapezius, respectively)

Myometric measurements were performed on each patient before and after the first, fourth and seventh treatments and 1 month after the last intervention in accordance with the manufacturer's instructions. The examiner carried out the measurements without knowing about the study group (blinding) and did not participate in the analysis of the obtained data.

IV (V) Assessment of health-related quality of life and pain sensation.

1. Assessment of health-related quality of life using the WHOQoL-BREF scale In order to compare the health-related quality of life before and after therapy, and 1 month after its completion, the subject completed the WHOQoL-BREF questionnaire. All required licenses for the use of the survey in the described research have been obtained.
2. Assessment of pain perception using the VAS scale Pain was assessed with the VAS analog pain scale in graphic form. The subjects were assessed on a scale of 1 to 10, immediately after the therapy of the muscles of the neck and shoulder girdle on days 1, 4 and 7. Patients were asked to answer: "How much did you feel pain in your muscles during the treatment?" The VAS scale also determined the intensity of the perceived headache during the last migraine attack before taking part in the treatment cycle and 1 month after the end of treatment by answering the question: "What was the intensity of the last headache / migraine episode?"

V. Statistical analysis. The test results were presented as the arithmetic mean (X) ± standard deviation (SD). The statistical analysis was performed using the STATISTICA v. 10 program (StatSoft, Inc. 2001, Kraków Poland). The Shapiro-Wilk test was used to check the normality of the distribution of serum concentrations of biochemical factors, biomechanical parameters, parameters of muscle properties, myometric tests, tests related to pain and health-related quality of life. Significant deviations from the normal distribution were found, so further analyzes were performed using non-parametric tests. In the case of the analysis of comparisons of several measurements (more than two), the Friedman ANOVA was used and when there were differences between the variables, the Post Hoc For Friedman test. For the comparative analysis of the two measurements (as in the case of the pain analysis), a non-parametric test was used for two dependent samples: Wilcoxon pairwise order. The results were considered statistically significant at the significance level of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

age: 18 to 65 years of age, female gender, migraine diagnosed by a specialist neurologist for at least 12 months, no metabolic, cardiological, neurological and orthopedic diseases within the shoulder girdle, and cervical spine, voluntary written consent for examination; criteria according to ICHD-3 allowing to classify the symptoms as migraines.

Exclusion Criteria:

minors or over 65 years of age, male gender, patients undergoing pharmacological treatment that cannot be discontinued; people with other headaches; past injuries of the musculoskeletal system in the cervical spine and shoulder girdle; skin diseases and other conditions such as deep vein thrombosis, osteoporosis; criteria for excluding migraine according to ICHD-3.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
ROM cervical spine | Before the first treatment.
  The measuring device allowed to assess the range of movement of the cervical spine with the motor control of the patient in the movement of the lateral to the right bend and left side, right and left rotations and forward bends. The ROM values will be expressed in degrees [°].
ROM cervical spine | After the first treatment.
  The measuring device allowed to assess the range of movement of the cervical spine with the motor control of the patient in the movement of the lateral to the right bend and left side, right and left rotations and forward bends. The ROM values will be expressed in degrees [°].
ROM cervical spine | Before the fourth treatment.
  The measuring device allowed to assess the range of movement of the cervical spine with the motor control of the patient in the movement of the lateral to the right bend and left side, right and left rotations and forward bends. The ROM values will be expressed in degrees [°].
ROM cervical spine | After the fourth treatment.
  The measuring device allowed to assess the range of movement of the cervical spine with the motor control of the patient in the movement of the lateral to the right bend and left side, right and left rotations and forward bends. The ROM values will be expressed in degrees [°].
ROM cervical spine | Before the seventh treatment.
  The measuring device allowed to assess the range of movement of the cervical spine with the motor control of the patient in the movement of the lateral to the right bend and left side, right and left rotations and forward bends. The ROM values will be expressed in degrees [°].
ROM cervical spine | After the seventh treatment.
  The measuring device allowed to assess the range of movement of the cervical spine with the motor control of the patient in the movement of the lateral to the right bend and left side, right and left rotations and forward bends. The ROM values will be expressed in degrees [°].
ROM cervical spine | Described data was collected for 1 month after the last intervention.
  The measuring device allowed to assess the range of movement of the cervical spine with the motor control of the patient in the movement of the lateral to the right bend and left side, right and left rotations and forward bends. The ROM values will be expressed in degrees [°].
Health-related quality of life | Before the first therapy.
  Health-related quality of life will be expressed as points of the WHOQoL-BREF scale [point]. The subject completed the WHOQoL-BREF questionnaire.
Health-related quality of life | After the first therapy.
  Health-related quality of life will be expressed as points of the WHOQoL-BREF scale [point]. The subject completed the WHOQoL-BREF questionnaire.
Health-related quality of life | 1 month after intervention completion, the subject completed the WHOQoL-BREF questionnaire again.
  Health-related quality of life will be expressed as points of the WHOQoL-BREF scale [point]. The subject completed the WHOQoL-BREF questionnaire.
Muscle pain perception | Day 1
  The subjects were assessed on a scale of 1 to 10 (VAS scale), immediately after the therapy of the muscles of the neck and shoulder girdle. Muscle pain perception will be expressed in [cm] as the distance between the two end points (between value 1 and 10) of visual analog scale.
Muscle pain perception | Day 4
  The subjects were assessed on a scale of 1 to 10 (VAS scale), immediately after the therapy of the muscles of the neck and shoulder girdle. Muscle pain perception will be expressed in [cm] as the distance between the two end points (between value 1 and 10) of visual analog scale.
Muscle pain perception | Day 7
  The subjects were assessed on a scale of 1 to 10 (VAS scale), immediately after the therapy of the muscles of the neck and shoulder girdle. Muscle pain perception will be expressed in [cm] as the distance between the two end points (between value 1 and 10) of visual analog scale.
Headache pain perception | Before the treatment cycle.
  The VAS scale also determined the intensity of the perceived headache during the last migraine attack. Headache pain perception will be expressed in [cm] as the distance between the two end points (between value 1 and 10) of visual analog scale (VAS).
Headache pain perception | 1 month after the end of treatment.
  The VAS scale also determined the intensity of the perceived headache during the last migraine attack. Headache pain perception will be expressed in [cm] as the distance between the two end points (between value 1 and 10) of visual analog scale (VAS).

SECONDARY OUTCOMES:
Myomentric parameter - Frequency | Before the first treatment.
  Frequency. Myotonometric frequency of natural oscillations (F-MYO) expressed in [Hz].
Myomentric parameter - Frequency | After the first treatment.
  Frequency. Myotonometric frequency of natural oscillations (F-MYO) expressed in [Hz].
Myomentric parameter - Frequency | Before the fourth treatment.
  Frequency. Myotonometric frequency of natural oscillations (F-MYO) expressed in [Hz].
Myomentric parameter - Frequency | After the fourth treatment.
  Frequency. Myotonometric frequency of natural oscillations (F-MYO) expressed in [Hz].
Myomentric parameter - Frequency | Before the seventh treatment.
  Frequency. Myotonometric frequency of natural oscillations (F-MYO) expressed in [Hz].
Myomentric parameter - Frequency | After the seventh treatment.
  Frequency. Myotonometric frequency of natural oscillations (F-MYO) expressed in [Hz].
Myomentric parameter - Frequency | 1 month after the last intervention.
  Frequency. Myotonometric frequency of natural oscillations (F-MYO) expressed in [Hz].
Myomentric parameter - Stiffness | Before the first treatment.
  Stiffness. Myotonometric stiffnes (S-MYO) expressed in [N/m].
Myomentric parameter - Stiffness | After the first treatment.
  Stiffness. Myotonometric stiffnes (S-MYO) expressed in [N/m].
Myomentric parameter - Stiffness | Before the fourth treatment.
  Stiffness. Myotonometric stiffnes (S-MYO) expressed in [N/m].
Myomentric parameter - Stiffness | After the fourth treatment.
  Stiffness. Myotonometric stiffnes (S-MYO) expressed in [N/m].
Myomentric parameter - Stiffness | Before the seventh treatment.
  Stiffness. Myotonometric stiffnes (S-MYO) expressed in [N/m].
Myomentric parameter - Stiffness | After the seventh treatment.
  Stiffness. Myotonometric stiffnes (S-MYO) expressed in [N/m].
Myomentric parameter - Stiffness | 1 month after the last intervention.
  Stiffness. Myotonometric stiffnes (S-MYO) expressed in [N/m].
Myomentric parameter - Decrement | Before the first treatment.
  Decrement. Myotonometric decrement of natural oscillations (D-MYO) expressed in logarithm of damping oscillations [log].
Myomentric parameter - Decrement | After the first treatment.
  Decrement. Myotonometric decrement of natural oscillations (D-MYO) expressed in logarithm of damping oscillations [log].
Myomentric parameter - Decrement | Before the fourth treatment.
  Decrement. Myotonometric decrement of natural oscillations (D-MYO) expressed in logarithm of damping oscillations [log].
Myomentric parameter - Decrement | After the fourth treatment.
  Decrement. Myotonometric decrement of natural oscillations (D-MYO) expressed in logarithm of damping oscillations [log].
Myomentric parameter - Decrement | Before the seventh treatment.
  Decrement. Myotonometric decrement of natural oscillations (D-MYO) expressed in logarithm of damping oscillations [log].
Myomentric parameter - Decrement | After the seventh treatment.
  Decrement. Myotonometric decrement of natural oscillations (D-MYO) expressed in logarithm of damping oscillations [log].
Myomentric parameter - Decrement | 1 month after the last intervention.
  Decrement. Myotonometric decrement of natural oscillations (D-MYO) expressed in logarithm of damping oscillations [log].
Blood parameter - SP | Before the treatment on the first day.
  The concentration of substance P was determined by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of substance P expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter - SP | After the treatment on the first day.
  The concentration of substance P was determined by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of substance P expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter - SP | 24 hours after the sixth treatment.
  The concentration of substance P was determined by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of substance P expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter S100beta | Before the treatment on the first day.
  The concentration of protein S100beta was determined by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of protein S100beta expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter S100beta | After the treatment on the first day.
  The concentration of protein S100beta was determined by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of protein S100beta expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter S100beta | 24 hours after the sixth treatment.
  The concentration of protein S100beta was determined by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of protein S100beta expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter CGRP | Before the treatment on the first day.
  The concentration of calcitonin gene-related peptide (CGRP) was determined by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of calcitonin gene-related peptide (CGRP) expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter CGRP | After the treatment on the first day.
  The concentration of calcitonin gene-related peptide (CGRP) was determined by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of calcitonin gene-related peptide (CGRP) expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter CGRP | 24 hours after the sixth treatment.
  The concentration of calcitonin gene-related peptide (CGRP) was determined by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of calcitonin gene-related peptide (CGRP) expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter BNDF | Before the treatment on the first day.
  The concentration of BNDF (brain-derived neurotrophic factor) was determied by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of BNDF expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter BNDF | After the treatment on the first day.
  The concentration of BNDF (brain-derived neurotrophic factor) was determied by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of BNDF expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.
Blood parameter BNDF | 24 hours after the sixth treatment.
  The concentration of BNDF (brain-derived neurotrophic factor) was determied by immunochemical ELISA method according to the kit manufacturers' instructions (R&D systems, London UK). The concentration of BNDF expressed in [ng/ml]. Peripheral blood from the ulnar vein was collected on an empty stomach between 6:00 am and 9:00 am into test tubes without serum anticoagulants.

CONTACTS AND LOCATIONS:
Overall Officials: Aneta Łuć, Study Director — Regional Research and Development Center in Biała Podlaska
Locations (1):
- Regional Research and Development Center, Biała Podlaska, Lublin Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adstrum S, Hedley G, Schleip R, Stecco C, Yucesoy CA. Defining the fascial system. J Bodyw Mov Ther. 2017 Jan;21(1):173-177. doi: 10.1016/j.jbmt.2016.11.003. Epub 2016 Nov 16. PMID 28167173
- [Background] Agostoni EC, Barbanti P, Calabresi P, Colombo B, Cortelli P, Frediani F, Geppetti P, Grazzi L, Leone M, Martelletti P, Pini LA, Prudenzano MP, Sarchielli P, Tedeschi G, Russo A; Italian chronic migraine group. Current and emerging evidence-based treatment options in chronic migraine: a narrative review. J Headache Pain. 2019 Aug 30;20(1):92. doi: 10.1186/s10194-019-1038-4. PMID 31470791
- [Background] Aird L, Samuel D, Stokes M. Quadriceps muscle tone, elasticity and stiffness in older males: reliability and symmetry using the MyotonPRO. Arch Gerontol Geriatr. 2012 Sep-Oct;55(2):e31-9. doi: 10.1016/j.archger.2012.03.005. Epub 2012 Apr 13. PMID 22503549
- [Background] Bengtsson A, Henriksson KG, Larsson J. Reduced high-energy phosphate levels in the painful muscles of patients with primary fibromyalgia. Arthritis Rheum. 1986 Jul;29(7):817-21. doi: 10.1002/art.1780290701. PMID 3741498
- [Background] Bizzini M, Mannion AF. Reliability of a new, hand-held device for assessing skeletal muscle stiffness. Clin Biomech (Bristol). 2003 Jun;18(5):459-61. doi: 10.1016/s0268-0033(03)00042-1. PMID 12763442
- [Background] Boska MD, Welch KM, Barker PB, Nelson JA, Schultz L. Contrasts in cortical magnesium, phospholipid and energy metabolism between migraine syndromes. Neurology. 2002 Apr 23;58(8):1227-33. doi: 10.1212/wnl.58.8.1227. PMID 11971091
- [Background] Bron C, Franssen J, Wensing M, Oostendorp RA. Interrater reliability of palpation of myofascial trigger points in three shoulder muscles. J Man Manip Ther. 2007;15(4):203-15. doi: 10.1179/106698107790819477. PMID 19066669
- [Background] Calandre EP, Hidalgo J, Garcia-Leiva JM, Rico-Villademoros F. Trigger point evaluation in migraine patients: an indication of peripheral sensitization linked to migraine predisposition? Eur J Neurol. 2006 Mar;13(3):244-9. doi: 10.1111/j.1468-1331.2006.01181.x. PMID 16618340
- [Background] Calandre EP, Hidalgo J, Garcia-Leiva JM, Rico-Villademoros F, Delgado-Rodriguez A. Myofascial trigger points in cluster headache patients: a case series. Head Face Med. 2008 Dec 30;4:32. doi: 10.1186/1746-160X-4-32. PMID 19116034
- [Background] Cernuda-Morollon E, Larrosa D, Ramon C, Vega J, Martinez-Camblor P, Pascual J. Interictal increase of CGRP levels in peripheral blood as a biomarker for chronic migraine. Neurology. 2013 Oct 1;81(14):1191-6. doi: 10.1212/WNL.0b013e3182a6cb72. Epub 2013 Aug 23. PMID 23975872
- [Background] Chaitow L, Fritz L. A Massage Therapist's Guide to Understanding, Locating and Treating Myofascial Trigger Points. Churchill Livingstone, Edinburgh 2006
- [Background] Chen Q, Basford J, An KN. Ability of magnetic resonance elastography to assess taut bands. Clin Biomech (Bristol). 2008 Jun;23(5):623-9. doi: 10.1016/j.clinbiomech.2007.12.002. Epub 2008 Feb 21. PMID 18206282
- [Background] Crooks DI, Newington K, Pilling L, Todd M. Assessing the feasibility of mobilisation of C0-C3 cervical segments to reduce headache in migraineurs. Int J Ther Reh 2018; 25(8): 382-394
- [Background] Dahlof C, Linde M. One-year prevalence of migraine in Sweden: a population-based study in adults. Cephalalgia. 2001 Jul;21(6):664-71. doi: 10.1046/j.1468-2982.2001.00218.x. PMID 11531898
- [Background] Dahlof CG, Dimenas E. Migraine patients experience poorer subjective well-being/quality of life even between attacks. Cephalalgia. 1995 Feb;15(1):31-6. doi: 10.1046/j.1468-2982.1995.1501031.x. PMID 7758095
- [Background] 21. Dejung B. Triggerpunkt-Therapie: Die Behandlungakuter Und chronischer Schmerzenim Bewegungsapparatmitmanueller Triggerpunkt-Therapie und Dry Needling. Berno, Hans Huber 2009; 13-37
- [Background] Diener HC, Bussone G, de Liano H, Eikermann A, Englert R, Floeter T, Gallai V, Gobel H, Hartung E, Jimenez MD, Lange R, Manzoni GC, Mueller-Schwefe G, Nappi G, Pinessi L, Prat J, Puca FM, Titus F, Voelker M; EMSASI Study Group. Placebo-controlled comparison of effervescent acetylsalicylic acid, sumatriptan and ibuprofen in the treatment of migraine attacks. Cephalalgia. 2004 Nov;24(11):947-54. doi: 10.1111/j.1468-2982.2004.00783.x. PMID 15482357
- [Background] Diener HC, Holle D, Dodick D. Treatment of chronic migraine. Curr Pain Headache Rep. 2011 Feb;15(1):64-9. doi: 10.1007/s11916-010-0159-x. PMID 21080112
- [Background] Edvinsson L. Calcitonin gene-related peptide (CGRP) and the pathophysiology of headache: therapeutic implications. CNS Drugs. 2001;15(10):745-53. doi: 10.2165/00023210-200115100-00001. PMID 11602001
- [Background] Espi-Lopez GV, Ruescas-Nicolau MA, Nova-Redondo C, Benitez-Martinez JC, Dugailly PM, Falla D. Effect of Soft Tissue Techniques on Headache Impact, Disability, and Quality of Life in Migraine Sufferers: A Pilot Study. J Altern Complement Med. 2018 Nov;24(11):1099-1107. doi: 10.1089/acm.2018.0048. Epub 2018 Apr 30. PMID 29708766
- [Background] Evans RW. Sports and Headaches. Headache. 2018 Mar;58(3):426-437. doi: 10.1111/head.13263. Epub 2018 Feb 5. PMID 29405284
- [Background] Evers S, Afra J, Frese A, Goadsby PJ, Linde M, May A, Sandor PS; European Federation of Neurological Societies. EFNS guideline on the drug treatment of migraine--revised report of an EFNS task force. Eur J Neurol. 2009 Sep;16(9):968-81. doi: 10.1111/j.1468-1331.2009.02748.x. PMID 19708964
- [Background] Amin FM, Aristeidou S, Baraldi C, Czapinska-Ciepiela EK, Ariadni DD, Di Lenola D, Fenech C, Kampouris K, Karagiorgis G, Braschinsky M, Linde M; European Headache Federation School of Advanced Studies (EHF-SAS). The association between migraine and physical exercise. J Headache Pain. 2018 Sep 10;19(1):83. doi: 10.1186/s10194-018-0902-y. PMID 30203180
- [Background] Farkkila M, Diener HC, Geraud G, Lainez M, Schoenen J, Harner N, Pilgrim A, Reuter U; COL MIG-202 study group. Efficacy and tolerability of lasmiditan, an oral 5-HT(1F) receptor agonist, for the acute treatment of migraine: a phase 2 randomised, placebo-controlled, parallel-group, dose-ranging study. Lancet Neurol. 2012 May;11(5):405-13. doi: 10.1016/S1474-4422(12)70047-9. Epub 2012 Mar 28. PMID 22459549
- [Background] Fernandez-de-Las-Penas C, Simons D, Cuadrado ML, Pareja J. The role of myofascial trigger points in musculoskeletal pain syndromes of the head and neck. Curr Pain Headache Rep. 2007 Oct;11(5):365-72. doi: 10.1007/s11916-007-0219-z. PMID 17894927
- [Background] Ferracini GN, Florencio LL, Dach F, Bevilaqua Grossi D, Palacios-Cena M, Ordas-Bandera C, Chaves TC, Speciali JG, Fernandez-de-Las-Penas C. Musculoskeletal disorders of the upper cervical spine in women with episodic or chronic migraine. Eur J Phys Rehabil Med. 2017 Jun;53(3):342-350. doi: 10.23736/S1973-9087.17.04393-3. Epub 2017 Jan 24. PMID 28118694
- [Background] Ferrari MD, Roon KI, Lipton RB, Goadsby PJ. Oral triptans (serotonin 5-HT(1B/1D) agonists) in acute migraine treatment: a meta-analysis of 53 trials. Lancet. 2001 Nov 17;358(9294):1668-75. doi: 10.1016/S0140-6736(01)06711-3. PMID 11728541
- [Background] Florencio LL, Ferracini GN, Chaves TC, Palacios-Cena M, Ordas-Bandera C, Speciali JG, Falla D, Grossi DB, Fernandez-de-Las-Penas C. Active Trigger Points in the Cervical Musculature Determine the Altered Activation of Superficial Neck and Extensor Muscles in Women With Migraine. Clin J Pain. 2017 Mar;33(3):238-245. doi: 10.1097/AJP.0000000000000390. PMID 27258994
- [Background] Gandolfi M, Geroin C, Vale N, Marchioretto F, Turrina A, Dimitrova E, Tamburin S, Serina A, Castellazzi P, Meschieri A, Ricard F, Saltuari L, Picelli A, Smania N. Does myofascial and trigger point treatment reduce pain and analgesic intake in patients undergoing onabotulinumtoxinA injection due to chronic intractable migraine? Eur J Phys Rehabil Med. 2018 Feb;54(1):1-12. doi: 10.23736/S1973-9087.17.04568-3. Epub 2017 Jul 27. PMID 28750504
- [Background] Ge HY, Fernandez-de-Las-Penas C, Yue SW. Myofascial trigger points: spontaneous electrical activity and its consequences for pain induction and propagation. Chin Med. 2011 Mar 25;6:13. doi: 10.1186/1749-8546-6-13. PMID 21439050
- [Background] Gerwin RD, Dommerholt J, Shah JP. An expansion of Simons' integrated hypothesis of trigger point formation. Curr Pain Headache Rep. 2004 Dec;8(6):468-75. doi: 10.1007/s11916-004-0069-x. PMID 15509461
- [Background] Glemser PA, Jaeger H, Nagel AM, Ziegler AE, Simons D, Schlemmer HP, Lehmann-Horn F, Jurkat-Rott K, Weber MA. 23Na MRI and myometry to compare eplerenone vs. glucocorticoid treatment in Duchenne dystrophy. Acta Myol. 2017 Mar;36(1):2-13. PMID 28690388
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Horwitz S, Stewart A. An Exploratory Study to Determine the Relationship between Cervical Dysfunction and Perimenstrual Migraines. Physiother Can. 2015 Winter;67(1):30-8. doi: 10.3138/ptc.2012-47. PMID 25931651
- [Background] Katsarava Z, Buse DC, Manack AN, Lipton RB. Defining the differences between episodic migraine and chronic migraine. Curr Pain Headache Rep. 2012 Feb;16(1):86-92. doi: 10.1007/s11916-011-0233-z. PMID 22083262
- [Background] Gozalov A, Jansen-Olesen I, Klaerke D, Olesen J. Role of BK(Ca) channels in cephalic vasodilation induced by CGRP, NO and transcranial electrical stimulation in the rat. Cephalalgia. 2007 Oct;27(10):1120-7. doi: 10.1111/j.1468-2982.2007.01409.x. Epub 2007 Aug 21. PMID 17714519
- [Background] Kollewe K, Escher CM, Wulff DU, Fathi D, Paracka L, Mohammadi B, Karst M, Dressler D. Long-term treatment of chronic migraine with OnabotulinumtoxinA: efficacy, quality of life and tolerability in a real-life setting. J Neural Transm (Vienna). 2016 May;123(5):533-40. doi: 10.1007/s00702-016-1539-0. Epub 2016 Mar 31. PMID 27032774
- [Background] Koppen H, van Veldhoven PL. Migraineurs with exercise-triggered attacks have a distinct migraine. J Headache Pain. 2013 Dec 21;14(1):99. doi: 10.1186/1129-2377-14-99. PMID 24359317
- [Background] Linde M. Migraine: a review and future directions for treatment. Acta Neurol Scand. 2006 Aug;114(2):71-83. doi: 10.1111/j.1600-0404.2006.00670.x. PMID 16867028
- [Background] Linton-Dahlof P, Linde M, Dahlof C. Withdrawal therapy improves chronic daily headache associated with long-term misuse of headache medication: a retrospective study. Cephalalgia. 2000 Sep;20(7):658-62. doi: 10.1111/j.1468-2982.2000.00099.x. PMID 11128824
- [Background] Lipton RB. Chronic migraine, classification, differential diagnosis, and epidemiology. Headache. 2011 Jul-Aug;51 Suppl 2:77-83. doi: 10.1111/j.1526-4610.2011.01954.x. PMID 21770929
- [Background] Lionetto L, Cipolla F, Guglielmetti M, Martelletti P. Fremanezumab for the prevention of chronic and episodic migraine. Drugs Today (Barc). 2019 Apr;55(4):265-276. doi: 10.1358/dot.2019.55.4.2970909. PMID 31050694
- [Background] Marusiak J, Jaskolska A, Koszewicz M, Budrewicz S, Jaskolski A. Myometry revealed medication-induced decrease in resting skeletal muscle stiffness in Parkinson's disease patients. Clin Biomech (Bristol). 2012 Jul;27(6):632-5. doi: 10.1016/j.clinbiomech.2012.02.001. Epub 2012 Feb 25. PMID 22365901
- [Background] Mualla B, Dilek B, Murat C, Nilgün I, Asuman G, Arsida B, İlknur A. The clinical efficiency of acupuncture in preventing migraine attacks and its effect on serotonin levels Turk J Phys Med Rehabil 2017; 63 (1): 59, 7
- [Background] Mueller-Wohlfahrt HW, Haensel L, Mithoefer K, Ekstrand J, English B, McNally S, Orchard J, van Dijk CN, Kerkhoffs GM, Schamasch P, Blottner D, Swaerd L, Goedhart E, Ueblacker P. Terminology and classification of muscle injuries in sport: the Munich consensus statement. Br J Sports Med. 2013 Apr;47(6):342-50. doi: 10.1136/bjsports-2012-091448. Epub 2012 Oct 18. PMID 23080315
- [Background] Myoton PRO For research use only: not for use in clinical, diagnostic or therapeutic procedures USER MANUAL, Londyn 2013; 25-26, 102-103.
- [Background] Ranoux D, Martine G, Espagne-Dubreuilh G, Amilhaud-Bordier M, Caire F, Magy L. OnabotulinumtoxinA injections in chronic migraine, targeted to sites of pericranial myofascial pain: an observational, open label, real-life cohort study. J Headache Pain. 2017 Dec;18(1):75. doi: 10.1186/s10194-017-0781-7. Epub 2017 Jul 21. PMID 28733943
- [Background] Song TJ, Cho SJ, Kim WJ, Yang KI, Yun CH, Chu MK. Sex Differences in Prevalence, Symptoms, Impact, and Psychiatric Comorbidities in Migraine and Probable Migraine: A Population-Based Study. Headache. 2019 Feb;59(2):215-223. doi: 10.1111/head.13470. Epub 2019 Jan 9. PMID 30623976
- [Background] Schroeter ML, Sacher J, Steiner J, Schoenknecht P, Mueller K. Serum S100B represents a new biomarker for mood disorders. Curr Drug Targets. 2013 Oct;14(11):1237-48. doi: 10.2174/13894501113149990014. PMID 23701298
- [Background] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849
- [Background] Shah JP, Danoff JV, Desai MJ, Parikh S, Nakamura LY, Phillips TM, Gerber LH. Biochemicals associated with pain and inflammation are elevated in sites near to and remote from active myofascial trigger points. Arch Phys Med Rehabil. 2008 Jan;89(1):16-23. doi: 10.1016/j.apmr.2007.10.018. PMID 18164325
- [Background] Simons D, Travell J. Myofascial Pain and Dysfunction The Trigger Point Manual - Vol. 1 - Upper Half of Body 1998
- [Background] Starling AJ, Vargas BB. A Narrative Review of Evidence-Based Preventive Options for Chronic Migraine. Curr Pain Headache Rep. 2015 Oct;19(10):49. doi: 10.1007/s11916-015-0521-0. PMID 26286071
- [Background] Stępień A. Treatment of primary headaches. Pain 2011; 12 (4): 7-10
- [Background] Sufrinko A, McAllister-Deitrick J, Elbin RJ, Collins MW, Kontos AP. Family History of Migraine Associated With Posttraumatic Migraine Symptoms Following Sport-Related Concussion. J Head Trauma Rehabil. 2018 Jan/Feb;33(1):7-14. doi: 10.1097/HTR.0000000000000315. PMID 28520665
- [Background] Tali D, Menahem I, Vered E, Kalichman L. Upper cervical mobility, posture and myofascial trigger points in subjects with episodic migraine: Case-control study. J Bodyw Mov Ther. 2014 Oct;18(4):569-75. doi: 10.1016/j.jbmt.2014.01.006. Epub 2014 Feb 6. PMID 25440209
- [Background] Terry DP, Huebschmann NA, Maxwell BA, Cook NE, Mannix R, Zafonte R, Seifert T, Berkner PD, Iverson GL. Preinjury Migraine History as a Risk Factor for Prolonged Return to School and Sports following Concussion. J Neurotrauma. 2019 Jan 1;36(1):142-151. doi: 10.1089/neu.2017.5443. Epub 2018 Aug 2. PMID 29732944
- [Background] Viir R, Laiho K, Kramarenko J, Mikkelsson M. Repeatability of trapezius muscle tone assessment by a myometric method. J Mech Med Biol 2006; 6: 215-228.
- [Background] Wells RE, Beuthin J, Granetzke L. Complementary and Integrative Medicine for Episodic Migraine: an Update of Evidence from the Last 3 Years. Curr Pain Headache Rep. 2019 Feb 21;23(2):10. doi: 10.1007/s11916-019-0750-8. PMID 30790138
- [Background] Zhang LM, Dong Z, Yu SY. Migraine in the era of precision medicine. Ann Transl Med. 2016 Mar;4(6):105. doi: 10.21037/atm.2016.03.13. PMID 27127758
- [Derived] Olesiejuk M, Chalimoniuk M, Sacewicz T. Myofascial trigger points therapy increases neck mobility and reduces headache pain in migraine patients - pilot study. BMC Musculoskelet Disord. 2025 Feb 1;26(1):105. doi: 10.1186/s12891-025-08360-1. PMID 39893364